CLINICAL TRIAL: NCT06500507
Title: Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Immunogenicity and Preliminary Effectiveness of QLS4131 Injection in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of QLS4131 in Patients With Recurrent or Refractory Multiple Myeloma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QLS4131-101
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Relapsed or Refractory Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QLS4131 (Experimental): Dose escalation and does expansion of QLS4131 injection will be evaluated.
  Interventions: Drug: QLS4131 Injection

INTERVENTIONS:
Drug: QLS4131 Injection — Participants confirming to the eligibility criteria will be assigned to 1 of the 9 dose groups (0.06/0.3/1 ~ 600 ug/kg, respectively) based on the sequence of inclusion.
  Other Names: A novel tri-specific humanized antibody

SUMMARY:
The purpose of this study is to characterize the safety of QLS4131 injection and to determine the recommended Phase 2 dose (RP2D) and to further evaluate the efficacy and safety of QLS4131 injection in participants with relapsed or refractory multiple myeloma at the recommended Phase 2 dose.

DETAILED DESCRIPTION:
Multiple myeloma (MM) is a malignant disease with abnormal proliferation of clonal plasma cell, which is often accompanied by multiple osteolytic damage, hypercalcemia, anemia, and kidney damage. QLS4131 is a novel tri-specific humanized antibody. The study consists 3 periods: screening phase, treatment phase and a post-treatment follow-up phase. The study will evaluate safety, tolerability, pharmacokinetics and preliminary antitumor activity of QLS4131 administered to participants with relapsed or refractory multiple myeloma. Total duration of study is up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, regardless of gender.
2. Subjects should be willing and able to comply with the study schedule and protocols.
3. Documented initial diagnosis of multiple myeloma according to International Myeloma Working Group (IMWG) diagnostic criteria.
4. Must have measurable disease as defined by the following: Serum M-protein greater than or equal to 1 g/dL; OR Urine M-protein greater than or equal to 200 mg/24 hours; OR Serum free light chain (FLC) assay; involved FLC level greater than or equal to 10 mg/dL provided the serum FLC ratio is abnormal.

Exclusion Criteria:

1. Known hypersensitivity to any of the ingredients of this product.
2. Known active central nervous system (CNS) involvement or exhibits clinical signs of meningeal involvement of multiple myeloma.
3. Has any active severe mental illness, medical illness, or other symptoms/conditions that may affect treatment, compliance, or the ability to provide informed consent, as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-08-30 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) | Approximately 2 years
  Determination of the recommended phase 2 dose (RP2D) of QLS41315 injection in patient with relapsed or refractory multiple myeloma
Incidence of adverse events（AEs） | Up to 2 years
  Assessing the incidence of adverse events (AEs) using the Common Terminology Criteria for Adverse Events (CTCAE Version 5).

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 2 years
  ORR assessed by the IMWG response criteria

CONTACTS AND LOCATIONS:
Overall Officials: Gang An, MD, Ph.D, Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No